CLINICAL TRIAL: NCT05689047
Title: Phase IIa Proof of Concept, Multicenter, Randomized, Open-label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of the Combination M5717 Plus Pyronaridine Administered Once Daily for 1 or 2 Days to Adults and Adolescents With Acute Uncomplicated Plasmodium Falciparum Malaria (CAPTURE 1)
Brief Title: Phase IIa Proof of Concept Study of M5717-Pyronaridine in Adults and Adolescents With Acute Uncomplicated Plasmodium Falciparum Malaria (CAPTURE 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201618_0033
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Acute Malaria
Keywords: M5717; Plasmodium mutants; Acute Malaria; Pyronaridine; Plasmodium falciparum; Polymerase chain reaction; Adequate Clinical and Parasitological Response; Plasmodium eukaryotic translation Elongation Factor 2
MeSH Terms: conditions — Acute malaria; Malaria, Falciparum | interventions — pyronaridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Safety Run-in Cohort M5717+Pyronaridine (Experimental): M5717 and pyronaridine once daily in a single day treatment regimen at low dose of 330 milligrams (mg) and 360 mg respectively.
  Interventions: Drug: M5717 330 mg; Drug: Pyronaridine 360 mg
- Part B: Dose escalation cohort; M5717+Pyronaridine (Experimental): After completion of Part A, if dose will be considered safe and well tolerated, the Internal Data Monitoring Committee (IDMC) will have the option to recommend dose adjustments. M5717 and pyronaridine once daily will be administered in an escalated dose in a single day or 2-day treatment regimen.
  Interventions: Drug: M5717 500 mg; Drug: M5717 660 mg; Drug: Pyronaridine 360 mg; Drug: Pyronaridine 540 mg; Drug: Pyronaridine 720 mg

INTERVENTIONS:
Drug: M5717 330 mg — Participants will receive orally 330 mg granules of M5717 in combination with pyronaridine dispersed in water under fasting condition.
  Arms: Part A: Safety Run-in Cohort M5717+Pyronaridine
Drug: M5717 500 mg — Adolescent participants with weight less than (<) 45 kilograms (kg) will receive orally 500 mg granules of M5717 in combination with pyronaridine dispersed in water once daily under fasting condition.
  Arms: Part B: Dose escalation cohort; M5717+Pyronaridine
Drug: M5717 660 mg — Adult and adolescent participants with weight more than or equal to (>=) 45 kg will receive orally 660 mg granules of M5717 in combination with pyronaridine dispersed in water once daily under fasting condition.
  Arms: Part B: Dose escalation cohort; M5717+Pyronaridine
Drug: Pyronaridine 360 mg — Participants will receive 360 mg of pyronaridine tablets in combination with M5717 under fasting condition.
  Arms: Part A: Safety Run-in Cohort M5717+Pyronaridine
Drug: Pyronaridine 360 mg — Participants with weight >=24 to <45 kg will receive 360 mg of tablets in combination with M5717 under fasting condition.
  Arms: Part B: Dose escalation cohort; M5717+Pyronaridine
Drug: Pyronaridine 540 mg — Participants with weight >=45 to <65 kg will receive 540 mg of Pyronaridine tablets in combination with M5717 under fasting condition.
  Arms: Part B: Dose escalation cohort; M5717+Pyronaridine
Drug: Pyronaridine 720 mg — Participants with weight >=65 kg will receive 720 mg of Pyronaridine tablets in combination with M5717 under fasting condition.
  Arms: Part B: Dose escalation cohort; M5717+Pyronaridine

SUMMARY:
The purpose of this study was to evaluate the safety, efficacy, and pharmacokinetic of the combination M5717 plus pyronaridine in participants with acute uncomplicated Plasmodium falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* Participants with microscopic confirmation of acute uncomplicated Plasmodium falciparum using Giemsa-stained thick and thin film
* P. falciparum parasitemia of 1,000 to 50,000 asexual parasites/microliter of blood in Part A and P. falciparum parasitemia of >1,000 to <= 150,000 asexual parasites/microliter of blood in Part B
* Axillary temperature >= 37.5 degree Celsius or tympanic temperature >= 38.0 degree Celsius (use as per Coronavirus disease 2019 (COVID-19) protocols at the site [only at Screening]), or history of fever during the previous 24 hours (at least documented verbally)
* The Investigator confirms that each participant agrees to use appropriate contraception and barriers, if applicable
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and this protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Mixed Plasmodium infections as per thin film microscopy results
* Signs and symptoms of severe malaria according to World Health Organisation (WHO) 2021 criteria (WHO 2021)
* Known liver abnormalities, liver cirrhosis (compensated or decompensated), known active or history of hepatitis B or C (testing not required), underlying hepatic injury or known severe liver disease, known gallbladder or bile duct disease, acute or chronic pancreatitis, or severe malnutrition
* Known history or evidence of clinically significant disorders such as, cardiovascular, respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological [including known Human Immunodeficiency Virus-Acquired Immunodeficiency Syndrome (HIV-AIDS)], neurological (including auditory), endocrine, infectious, malignancy, psychiatric, history of convulsions, or other abnormality (including head trauma)
* Previous treatment with pyronaridine as part of a combination therapy during the last 3 months
* Prior antimalarial therapy or antibiotics with antimalarial activity within a minimum of their 5 plasma half-lives (or within 4 weeks of Screening if half-life is unknown)
* Participants taking medications prohibited by the protocol
* Other protocol defined exclusion criteria could apply

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (5):
- Burkina Faso (2):
  - Institut de Recherche en Sciences de la Santé (IRSS), Nanoro
  - Groupe de Recherche Action en Santé (GRAS), Ouagadougou
- Centre de Recherches Médicales de Lambaréné (CERMEL), Lambaréné, Gabon
- Centro de Investigação em saúde de Manhiça/Fundação Manhiça (CISM/FM), Maputo, Mozambique
- Infectious Diseases Research Collaboration (IDRC), Tororo, Uganda

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201618_0033
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on the data evaluated in Cohort A and Cohort B0, it was decided not to conduct Cohorts B1, B2 and B3 and study was completed after completion of Cohorts A and B0. Therefore, no enrollment was done in Cohorts B1, B2, and B3. All study analyses were conducted using data from Cohort A and B0 only.
Groups:
- Cohort A: M5717+Pyronaridine: Participants received 330 milligrams (mg) granules of M5717 orally in combination with 360 mg pyronaridine tablet
- Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine: Participants with weight less than (<) 45 kilograms (kg) received 500 mg granules of M5717 orally in combination with 360 mg pyronaridine daily or adult and adolescent participants with weight more than or equal to (>=) 45 kg received orally 660 mg granules of M5717 in combination with 540 mg pyronaridine once daily under fasting condition. Participants with weight >=65 kg received 720 mg of Pyronaridine tablets in combination with M5717 under fasting condition. The follow up period for participants was 28 days.
Period: Overall Study
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Started | 12 | 26
Completed | 11 | 25
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine | Total
Number analyzed (Participants) | 12 | 26 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23 (9.56) | 18 (9.03) | 20 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 1 | 11 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Hispanic or Latino | 0 | 1 | 1
  Ethnicity-Not Hispanic or Latino | 0 | 25 | 25
  Ethnicity-Unknown or Not Reported | 12 | 0 | 12
  Race-Black or African American | 12 | 25 | 37
  Race-White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and Related TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant. TEAEs are defined as AEs which started at or after the administration of study intervention (study treatment) or which started prior to the first administration of study intervention but worsened after the dose intake, until the last scheduled assessment will be regarded as treatment-emergent, but before established rescue antimalarial treatment is administered, if required. A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. A TEAE was considered to be "related" if a causal relationship between study treatment and the TEAE is at least reasonably possible.
Time Frame: Day 1 up to Day 43
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: M5717+Pyronaridine
Number analyzed (Participants) | 12
Participants
  TEAEs | 9
  Serious TEAEs | 0
  Related TEAEs | 1

2. Primary Outcome: Cohort A: Number of Participants With Clinically Significant Change From Baseline in Safety Laboratory Parameters
Description: Number of participants with clinically significant change from baseline in laboratory parameters were reported. Clinical Significance was decided by the investigator. Laboratory investigation included hematology, biochemistry, and coagulation.
Time Frame: Day 1 up to Day 29
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: M5717+Pyronaridine
Number analyzed (Participants) | 12
Participants | 0

3. Primary Outcome: Cohort A: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings
Description: Number of participants with clinically significant change from baseline in ECG parameters were reported. Clinical Significance was decided by the investigator. The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. The parameters included heart rate (HR), Respiratory Rate, Pulse Rate, QRS, QT and QTcB calculated by the Bazett formula.
Time Frame: Day 1 up to Day 29
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: M5717+Pyronaridine
Number analyzed (Participants) | 12
Participants | 0

4. Primary Outcome: Cohort A: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Number of participants with clinically significant change from baseline in vital signs. Clinical Significance was decided by the investigator. Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate.
Time Frame: Day 1 up to Day 29
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: M5717+Pyronaridine
Number analyzed (Participants) | 12
Participants | 0

5. Primary Outcome: Cohort B0: Percentage of Participants With Polymerase Chain Reaction (PCR)-Adjusted Adequate Clinical and Parasitological Response (ACPR)
Description: PCR-adjusted ACPR 28 days after first treatment (i.e., on Day 29) was defined as absence of parasitemia (thick smear/microscopy, after adjustment for parasitemia due to new infections as determined by genotyping using PCR techniques), irrespective of axillary temperature, in participants who did not previously meet any of the criteria of Early treatment failure (ETF), Late clinical failure (LCF), or Late parasitological failure (LPF).
Time Frame: At Day 29
Population: The Full Analysis Set included all enrolled participants. ACPR could not be assessed for 1 participant due to missing parasites assessment at Day 28. Here "Number Analyzed" is equivalent to the number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 24
percentage of participants | 92.3 [75.9 to 97.9]

6. Secondary Outcome: Cohort A and Cohort B0: Area Under Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M5717 and Pyronaridine
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination. Calculated as AUC0-inf = AUC0-tlast + Clast pred/ lambda z.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: The Pharmacokinetics (PK) analysis set included all participants, who received more than equal to 1 dose of study intervention, have no clinically important protocol deviations or important events affecting PK and provide more than equal to (>=) 1 measurable post-dose concentration. Dose wise results have been reported for M5717 and Pyronaridine as per the planned analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter(h*ng/ml)
Groups:
- Cohort A: M5717 330 mg: Participants received 330 milligrams (mg) granules of M5717 orally.
- Cohort B0: M5717 500 mg: Participants with weight less than (<) 45 kilograms (kg) received 500 mg granules of M5717 orally.
- Cohort B0: M5717 660 mg: Adult and adolescent participants with weight more than or equal to (>=) 45 kg received orally 660 mg granules of M5717.
- Cohort A and B0: Pyronaridine 360 mg: Participants received 360 mg of pyronaridine tablets under fasting conditions.
- Cohort B0: Pyronaridine 540 mg: Participants with weight >=45 to <65 kg received 540 mg of Pyronaridine tablets under fasting conditions.
- Cohort B0: Pyronaridine 720 mg: Participants with weight >=65 kg received 720 mg of Pyronaridine tablets under fasting conditions.
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
hour*nanogram/milliliter(h*ng/ml) | 11194.723 (0.238) | 33307.278 (0.153) | 33756.087 (0.384) | 4397.819 (0.590) | 8557.596 (0.347) | 5899.378 (0.289)

7. Secondary Outcome: Cohort A and Cohort B0: Area Under Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24) of M5717 and Pyronaridine
Description: The AUC from time zero (dosing time) to 24 hours post dose was calculated using the mixed log linear trapezoidal rule (linear up, log down) using the nominal dosing interval.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: The PK analysis set included all participants, who received more than equal to 1 dose of study intervention, have no clinically important protocol deviations or important events affecting PK and provide >= 1 measurable post-dose concentration. Dose wise results have been reported for M5717 and Pyronaridine as per the planned analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
h*ng/ml | 3663.092 (0.373) | 13063.782 (0.127) | 12038.002 (0.393) | 1206.579 (0.417) | 2113.426 (0.399) | 1603.917 (0.197)

8. Secondary Outcome: Cohort A and Cohort B0: Area Under Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-tlast) of M5717 and Pyronaridine
Description: The AUC from time zero (= dosing time) to the time of the last quantifiable concentration (tlast), calculated using the mixed log linear trapezoidal rule (linear up, log down)
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
h*ng/ml | 9877.195 (0.455) | 32747.057 (0.153) | 33275.071 (0.391) | 4397.819 (0.590) | 8557.596 (0.347) | 5899.378 (0.289)

9. Secondary Outcome: Cohort A and Cohort B0: Apparent Total Clearance (CL/F) of M5717 and Pyronaridine
Description: The apparent total body clearance of study intervention following extravascular administration. CL/ F was calculated by oral dose divided by Area under the plasma concentration curve 0- infinity.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (l/h)
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
Liters/hour (l/h) | 29.478 (0.238) | 15.012 (0.153) | 19.552 (0.384) | 81.859 (0.590) | 63.102 (0.347) | 122.047 (0.289)

10. Secondary Outcome: Cohort A and Cohort B0: Maximum Plasma Concentration (Cmax) of M5717 and Pyronaridine
Description: Cmax was taken directly from the observed concentration-time curve.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
ng/ml | 269.358 (0.483) | 956.145 (0.173) | 991.144 (0.385) | 125.600 (44.565) | 191.000 (78.773) | 138.000 (15.122)

11. Secondary Outcome: Cohort A and Cohort B0: Apparent Terminal Half-Life of M5717 and Pyronaridine
Description: t1/2 was the time measured for the concentration to decrease by one half. t1/2 was calculated by natural log 2 divided by Lambda z.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
hours (h) | 74.523 (0.264) | 65.638 (0.152) | 84.202 (0.325) | 174.918 (0.599) | 228.509 (0.233) | 229.264 (0.314)

12. Secondary Outcome: Cohort A and Cohort B0: Time to Reach Maximum Plasma Concentration (Tmax) of M5717 and Pyronaridine
Description: tmax was obtained directly from the concentration versus time curve.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
hours | 3.179 (0.480) | 2.784 (0.385) | 3.196 (0.508) | 2.778 (0.325) | 3.394 (0.599) | 4.444 (0.767)

13. Secondary Outcome: Cohort A and Cohort B0: Apparent Volume of Distribution (Vz/F) of M5717 and Pyronaridine
Description: The apparent volume of distribution during the terminal phase following extravascular administration. Vz/F = Dose/(AUC0-∞*λz) following single dose.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (l)
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
liters (l) | 3169.306 (0.389) | 1421.536 (0.220) | 2375.135 (0.647) | 20657.284 (0.459) | 20802.718 (0.250) | 40368.007 (0.224)

14. Secondary Outcome: Cohort A and Cohort B0: Dose Normalized Area Under the Curve From Time Zero to 24 Hours Post Dose (AUC0-24h/Dose) of M5717 and Pyronaridine
Description: The dose normalized AUC from time zero to 24 hours post dose. Normalized using the dose, using the formula AUC0-24/Dose.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
h*ng/mL/mg | 11.100 (0.373) | 26.128 (0.127) | 18.239 (0.393) | 3.352 (0.417) | 3.914 (0.399) | 2.228 (0.197)

15. Secondary Outcome: Cohort A and Cohort B0: Dose Normalized Area Under the Curve From Time Zero to the Last Sampling Time (AUC0-tlast/Dose) of M5717 and Pyronaridine
Description: The dose normalized AUC from time zero to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Normalized using the dose, using the formula AUC0-tlast /Dose.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
h*ng/mL/mg | 29.931 (0.455) | 65.494 (0.153) | 50.417 (0.391) | 11.033 (0.625) | 14.792 (0.366) | 7.639 (0.303)

16. Secondary Outcome: Cohort A and Cohort B0: Dose Normalized Area Under the Curve From Time Zero Extrapolated to Infinity (AUC0-∞/Dose) of M5717 and Pyronaridine
Description: The dose normalized AUC from time zero extrapolated to infinity. Normalized using dose, using the formula AUC0-∞ /Dose.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
h*ng/mL/mg | 33.923 (0.238) | 66.615 (0.153) | 51.146 (0.384) | 12.216 (0.590) | 15.847 (0.347) | 8.194 (0.289)

17. Secondary Outcome: Cohort A and Cohort B0: Terminal Elimination Rate Constant (Lambda z) of M5717 and Pyronaridine
Description: Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
hours (h) | 0.009 (0.264) | 0.011 (0.152) | 0.008 (0.325) | 0.004 (0.599) | 0.003 (0.233) | 0.003 (0.314)

18. Secondary Outcome: Cohort A and Cohort B0: Dose Normalized Maximum Concentration (Cmax/Dose) of M5717 and Pyronaridine
Description: The dose normalized maximum concentration. Normalized using the dose, and the formula Cmax /Dose.
Time Frame: Predose and Post dose on Day 1, Post dose on Day 2, 3, 4, 8, 15, 22, 29 and Day 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Cohort A: M5717 330 mg | Cohort B0: M5717 500 mg | Cohort B0: M5717 660 mg | Cohort A and B0: Pyronaridine 360 mg | Cohort B0: Pyronaridine 540 mg | Cohort B0: Pyronaridine 720 mg
Number analyzed (Participants) | 12 | 9 | 15 | 21 | 11 | 4
ng/mL/mg | 0.816 (0.483) | 1.912 (0.173) | 1.502 (0.385) | 12.216 (0.590) | 15.847 (0.347) | 8.194 (0.289)

19. Secondary Outcome: Cohort A and Cohort B0: Percentage of Participants With Early Treatment Failure (ETF)
Description: Early treatment failure (ETF) was defined as meeting any of the following : 1. Danger signs or severe malaria 1, 2, or 3 days after treatment, in the presence of parasitemia2. Parasitemia 2 days after treatment higher than on day of treatment, irrespective of axillary temperature
  • Parasitemia 3 days after treatment with temperature ≥ 37.5°C 3. Parasitemia 3 days after treatment ≥ 25% of count on day of treatment. ETF rate will be estimated with 95% confidence intervals. Confidence intervals was derived by use of Wilson's score method.
Time Frame: Up to Day 3 post treatment on Day 1
Population: The Full Analysis Set (FAS) included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 12 | 26
percentage of participants | 0.0 [0.0 to 24.3] | 0.0 [0.0 to 12.9]

20. Secondary Outcome: Cohort A and Cohort B0: Percentage of Participants With Late Clinical Failure (LCF)
Description: Late clinical failure (LCF) was defined as:1. Danger signs or severe malaria in the presence of parasitemia on any day between 4 and 28 days after treatment (i.e., between Days 5 and 29) in participants who did not previously meet any of the criteria of ETF. 2. Presence of parasitemia on any day between 4 and 28 days after treatment with temperature ≥ 37.5°C in participants who did not previously meet any of the criteria of ETF. LCF was estimated with 95% confidence intervals. Confidence intervals will be derived by use of Wilson's score method.
Time Frame: Day 1 up to Day 29
Population: The FAS included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 12 | 26
percentage of participants | 0.0 [0.0 to 24.3] | 0.0 [0.0 to 12.9]

21. Secondary Outcome: Cohort A and Cohort B0: Percentage of Participants With Late Parasitological Failure (LPF)
Description: Late parasitological failure (LPF) was defined as: Presence of parasitemia on any day between 7 and 28 days after treatment (i.e., between Days 8 and 29) with temperature < 37.5°C in participants who did not previously meet any of the criteria of ETF or LCF. LPF was estimated with 95% confidence intervals. Confidence intervals will be derived by use of Wilson's score method.
Time Frame: From Day 8 to Day 29
Population: The FAS included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 12 | 26
percentage of participants | 0.0 [0.0 to 24.3] | 0.0 [0.0 to 12.9]

22. Secondary Outcome: Cohort A: Percentage of Participants With Polymerase Chain Reaction (PCR)-Adjusted Adequate Clinical and Parasitological Response (ACPR)
Description: PCR-adjusted ACPR 28 and 42 days after treatment defined as absence of parasitemia (thick smear/microscopy, after adjustment for parasitemia due to new infections as determined by genotyping using PCR techniques), irrespective of axillary temperature, in participants who did not previously meet any of the criteria of ETF, LCF, or LPF.
Time Frame: Day 28 and 42
Population: The FAS included all enrolled participants. ACPR could not be assessed for 1 patient due to missing parasites assessment at Day 28.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: M5717+Pyronaridine
Number analyzed (Participants) | 12
percentage of participants
  Day 28 | 91.7 [64.6 to 98.5]
  Day 42 | 91.7 [64.6 to 98.5]

23. Secondary Outcome: Cohort A and B0: Percentage of Participants With Crude Adequate Clinical and Parasitological Response (ACPR)
Description: Crude ACPR 28 and 42 days after first dose is defined as absence of parasitemia (parasite count = 0) from thick smear/microscopy, irrespective of axillary temperature, in participants who did not previously meet any of the criteria of ETF, LCF, or LPF.
Time Frame: Day 28 and 42
Population: The FAS included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 12 | 26
percentage of participants
  Day 28 | 91.7 [64.6 to 98.5] | 92.3 [75.9 to 97.9]
  Day 42 | 91.7 [64.6 to 98.5] | 76.9 [57.9 to 89.0]

24. Secondary Outcome: Cohort A and Cohort B0: Time to Fever Clearance as Estimated by Kaplan-Meier Method
Description: Fever clearance time was defined as the time from first dosing to the first measurement of temperature < 37.5°C for 2 consecutive temperature readings plus confirmed normal temperature 24 h after the first normal body temperature reading. This analysis was done on participants with fever.
Time Frame: Day 1 up to Day 29
Population: The FAS included all enrolled participants. Here "Number Analyzed" is equivalent to the number of participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 1 | 9
hours | 6.0 [6.0 to 6.0] | 6.2 [6.0 to 17.9]

25. Secondary Outcome: Cohort A and Cohort B0: Parasite Clearance Time as Estimated by Kaplan-Meier Method
Description: Parasite clearance time defined as time from dosing to the first negative (no parasites) film
Time Frame: Day 1 up to Day 43
Population: The FAS included all enrolled participants.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 12 | 26
days | 4.0 [3.0 to 9.0] | 4.5 [2.0 to 10.0]

26. Secondary Outcome: Cohort B0: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and Related TEAEs
Description: as for outcome 1
Time Frame: Day 1 up to Day 43
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
Number analyzed (Participants) | 26
Participants
  TEAEs | 16
  Serious TEAEs | 0
  Related TEAEs | 0

ADVERSE EVENTS:
Time Frame: Up to Day 43
Arm/Group | Cohort A: M5717+Pyronaridine | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/26
Other Adverse Events (participants affected / at risk) | 9/12 | 16/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: M5717+Pyronaridine (N=12) | Cohort B0: Dose Escalation Cohort: M5717+Pyronaridine (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 2 (2)
Malaria (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 5 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT05689047/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT05689047/SAP_001.pdf